CLINICAL TRIAL: NCT00411554
Title: Sitagliptin (MK0431) Phase III Double-blind Comparative Study - Type 2 Diabetes Mellitus -
Brief Title: A Study of Sitagliptin in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Diet/Exercise Therapy (0431-054)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-054; 2006_051
Record Dates: First submitted 2006-12-13; First posted 2006-12-14 (Estimated); Results first posted 2009-09-25 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; voglibose

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Sitagliptin 50 mg QD (Experimental): sitagliptin 50 mg orally once daily (QD=once daily)
  Interventions: Drug: sitagliptin phosphate
- Voglibose 0.2 mg TID (Active Comparator): voglibose 0.2 mg orally three times daily (TID= three times daily)
  Interventions: Drug: Comparator: voglibose

INTERVENTIONS:
Drug: sitagliptin phosphate — sitagliptin 50 mg orally once daily QD. Duration of Treatment: 12 Weeks
  Other Names: MK0431
  Arms: Sitagliptin 50 mg QD
Drug: Comparator: voglibose — voglibose 0.2 mg orally three times daily TID. Duration of Treatment: 12 Weeks
  Other Names: voglibose
  Arms: Voglibose 0.2 mg TID

SUMMARY:
The clinical study determines the safety and efficacy of Sitagliptin (MK0431) in patients with type 2 diabetes mellitus who have inadequate glycemic control on diet/exercise therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients have type 2 diabetes mellitus on diet/exercise therapy

Exclusion Criteria:

* Patients have type 1 diabetes mellitus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2007-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Iwamoto Y, Tajima N, Kadowaki T, Nonaka K, Taniguchi T, Nishii M, Arjona Ferreira JC, Amatruda JM. Efficacy and safety of sitagliptin monotherapy compared with voglibose in Japanese patients with type 2 diabetes: a randomized, double-blind trial. Diabetes Obes Metab. 2010 Jul;12(7):613-22. doi: 10.1111/j.1463-1326.2010.01197.x. PMID 20590736

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III.
  First patient in: 6 January 2007. Last patient, last visit: 15 August 2007.
  The study was conducted at 71 centers in Japan.
Pre-assignment Details: Patients at least 20 years of age with type 2 diabetes mellitus and inadequate glycemic control (HbA1c ≥6.5% and <10% at Week -2) were eligible for randomization following at least 8 weeks of diet/exercise and antihyperglycemic agent (AHA) wash-off (for patients previously on an AHA), including a 2-week placebo run-in.
Groups:
- Sitagliptin 50 mg QD: The Sitagliptin group includes data from all patients randomized to receive treatment with sitagliptin 50 mg orally once daily (QD=once daily).
- Voglibose 0.2 mg TID: The Voglibose group includes data from all patients randomized to receive treatment with voglibose 0.2 mg orally three times daily (TID= three times daily).
Period: Overall Study
Arm/Group | Sitagliptin 50 mg QD | Voglibose 0.2 mg TID
Started | 163 (Study enrolled slightly more than the target of N=155) | 156 (Study enrolled slightly more than the target of N=155)
Completed | 155 | 147
Not Completed | 8 | 9
Not completed — Adverse Event | 2 | 4
Not completed — Lack of Efficacy | 2 | 5
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Patient Moved | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 50 mg QD | Voglibose 0.2 mg TID | Total
Number analyzed (Participants) | 163 | 156 | 319
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (10.1) | 60.6 (10.0) | 60.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 62 | 107
  Male | 118 | 94 | 212
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 148.7 (34.2) | 148.9 (31.0) | 148.8 (32.6)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percent] | 7.8 (0.9) | 7.8 (0.9) | 7.8 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 12
Description: HbA1c is measured as a percent. Thus, this change from baseline reflects the Week 12 HbA1c percent minus the Week 0 HbA1c percent.
Time Frame: Baseline and Week 12
Population: The Per Protocol Population included patients with baseline and Week 12 (i.e., final primary timepoint) values for this outcome and excluded patients who met predefined criteria for major protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 155 | 146
Percent | -0.70 [-0.78 to -0.62] | -0.30 [-0.39 to -0.22]
Statistical Analysis 1: Comparison: Sitagliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Non-Inferiority or Equivalence — Non-inferiority margin (Sitagliptin minus Voglibose) = 0.2 percent; p < 0.001, ANCOVA — This p-value corresponds to a test of superiority that was performed after success was achieved in the test of non-inferiority (reported under "Estimation" below), according to the pre-specified analysis plan; ANCOVA model with terms of treatment, prior antihyperglycemic medication status and baseline was used to compare two groups; Least-squares Mean Difference = -0.39, 95% CI [-0.51 to -0.28] — ANCOVA model with terms of treatment, prior antihyperglycemic medication status and baseline was used to show non-inferiority and superiority to voglibose (closed procedure) and to estimate difference of two groups and its 95% confidence interval

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 12
Description: Change from baseline at Week 12 is defined as fasting plasma glucose at Week 12 minus fasting plasma glucose at Week 0.
Time Frame: Baseline and Week 12
Population: The Per Protocol Population included patients with baseline and Week 12 (i.e., final primary timepoint) values for this outcome and excluded patients who met predefined criteria for protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 155 | 146
mg/dL | -19.6 [-22.8 to -16.4] | -8.9 [-12.2 to -5.5]
Statistical Analysis 1: Comparison: Sitagliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least-squares Mean Difference = -10.7, 95% CI [-15.3 to -6.2] — ANCOVA model with terms of treatment, prior antihyperglycemic medication status and baseline was used to show superiority to voglibose and to estimate difference of two groups and its 95% confidence interval

3. Secondary Outcome: Change From Baseline in 2 Hour Postprandial Glucose at Week 12
Description: Change from baseline at Week 12 is defined as 2-hour postprandial glucose Week 12 minus 2-hour postprandial glucose Week 0.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 50 mg QD | Voglibose 0.2 mg TID
Number analyzed (Participants) | 152 | 146
mg/dL | -51.0 [-56.5 to -45.4] | -32.2 [-37.9 to -26.5]
Statistical Analysis 1: Comparison: Sitagliptin 50 mg QD vs Voglibose 0.2 mg TID; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least-squares Mean Difference = -18.8, 95% CI [-26.7 to -10.9] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Arm/Group | Sitagliptin 50 mg QD | Voglibose 0.2 mg TID
Serious Adverse Events (participants affected / at risk) | 1 | 2
Other Adverse Events (participants affected / at risk) | 32 | 62
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Sitagliptin 50 mg QD | Voglibose 0.2 mg TID
Cellulitis (Infections and infestations) | 1/163 | 0/156
Foot fracture (Injury, poisoning and procedural complications) | 0/163 | 1/156
Crohn's disease (Gastrointestinal disorders) | 0/163 | 1/156
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Sitagliptin 50 mg QD | Voglibose 0.2 mg TID
Abdominal distension (Gastrointestinal disorders) | 7/163 | 14/156
Diarrhoea (Gastrointestinal disorders) | 4/163 | 12/156
Flatulence (Gastrointestinal disorders) | 7/163 | 17/156
Nasopharyngitis (Infections and infestations) | 22/163 | 24/156
Alanine aminotransferase increased (Investigations) | 1/163 | 11/155

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.